CLINICAL TRIAL: NCT04597502
Title: "The Effects of Synastol TC (Standardized Terminalia Chebula Fruit Extract) on the Gut Microbiome and Skin Biophysical Properties"
Brief Title: The Effects of Terminalia Chebula Fruit Extract on the Gut Microbiome and Skin Biophysical Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Sytheon Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TC-0203
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Human Microbiome
Keywords: gut microbiome; skin; dermatology; terminalia chebula
MeSH Terms: interventions — chebulae fruit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral Placebo, Topical Placebo (Placebo Comparator): Oral Placebo, Topical Placebo on both forearms and dorsal hands
  Interventions: Dietary Supplement: Placebo; Other: Topical Placebo
- Oral Placebo, Topical TC (Experimental): Oral Placebo, Topical TC on both forearms and dorsal hands
  Interventions: Dietary Supplement: Placebo; Other: Topical Terminalia Chebula
- Oral TC, Topical Placebo (Experimental): Oral TC, Topical Placebo on both forearms and dorsal hands
  Interventions: Dietary Supplement: Terminalia Chebula fruit extract; Other: Topical Placebo
- Oral TC, Topical TC (Experimental): Oral TC, Topical TC on both forearms and dorsal hands
  Interventions: Dietary Supplement: Terminalia Chebula fruit extract; Other: Topical Terminalia Chebula

INTERVENTIONS:
Dietary Supplement: Terminalia Chebula fruit extract — Oral TC fruit extract supplement taken by mouth twice per day
  Arms: Oral TC, Topical Placebo; Oral TC, Topical TC
Dietary Supplement: Placebo — Oral placebo taken by mouth twice per day
  Arms: Oral Placebo, Topical Placebo; Oral Placebo, Topical TC
Other: Topical Terminalia Chebula — Applied to both forearms and dorsal hands
  Arms: Oral Placebo, Topical TC; Oral TC, Topical TC
Other: Topical Placebo — Applied to both forearms and dorsal hands
  Arms: Oral Placebo, Topical Placebo; Oral TC, Topical Placebo

SUMMARY:
The purpose of this study is to assess the use of oral Terminalia chebula fruit extract on the gut microbiome and skin biophysical properties. The fruit is commonly used for skin treatments in India. It is thought to have antioxidant properties, reduce inflammation and affect the microorganisms in the gut.

The information the investigators will learn from this study may indicate how and if oral dosing can affect the skin and gut microbiome. This may lead to an improved understanding of the skin and determine whether these oral products are effective for improving the skin's appearance.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 25 to 55 years of age
2. Subject must be able to read and comprehend study procedures and consent forms.
3. BMI 25-35

Exclusion Criteria:

1. Subjects must have no history of malignancy, kidney disease, or chronic steroid use.
2. No history of smoking or chewing tobacco or vaping nicotine based products within the past year or if the pack-year history of smoking tobacco is greater than 5 pack-years.
3. No history of anorexia
4. Those that are currently taking serotonin or SSRIs.
5. No intake of pomegranate containing drinks, walnuts, and strawberries two weeks prior to enrollment and throughout the study
6. Those who are unable to discontinue topical medications for two weeks.
7. Individuals who have had any medical or cosmetic procedure, such as laser resurfacing, or plastic surgery to the test site (face) within the last 6 months. This includes botulinum toxin, dermal fillers, collagen or other similar cosmetic procedure
8. Individuals who are currently using or during the past 30 days have used hydroquinone, or a retinoid such as Retin A, or other Rx/OTC Retinoid, or steroids.
9. Those who are unable to discontinue systemic antibiotics or oral probiotics for one month prior starting the study.
10. Those who are unable to discontinue their Triphala or Terminalia chebula regimen for one month prior to starting study.
11. Subjects who are postmenopausal or perimenopausal as determined by the investigator based on history or documented menopause
12. Males will be excluded to reduce the contribution from gender-based differences in testosterone which can affect sebum production on the face.
13. Those who are pregnant or breastfeeding
14. Those that are prisoners or cognitively impaired
15. Those who have a known allergy to Triphala or Terminalia chebula

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Stool microbiome diversity | 8 weeks
  Stool is collected and analyzed for species of bacteria through nucleic acid sequencing.
Sebum production | 8 weeks
  Delfin Sebumeter: 0-150 micrograms/cm^2

SECONDARY OUTCOMES:
Transepidermal water loss | 8 weeks
  Delfin Vapometer 0-300g/m^2h
Facial pigmentation | 8 weeks
  SkinColorCatchRGB range: 25-246 per channel
Facial redness - Device Based | 8 weeks
  SkinColorCatch colorimeter RGB range: 25-246 per channel
Facial wrinkles | 8 weeks
  BTBP Clarity Mini 3D camera: Wrinkle severity (depth and width measurement in unitless units)
Facial shine | 8 weeks
  BTBP Clarity Mini 3D: (Surface reflection measured in unitless units)
hand and arm pigmentation | 8 weeks
  SkinColorCatch colorimeter RGB range: 25-246 per channel
hand and arm redness | 8 weeks
  SkinColorCatch colorimeter RGB range: 25-246 per channel
Tolerability of Topical Products | 8 weeks
  Subjective Tolerability Questionnaire is collected
Skin typing questionnaire | 8 weeks
  Subjective Questionnaire is collected
Ayurvedic typing questionnaire | 8 weeks
  Subjective Questionnaire is collected
Salivary diurnal cortisol slope | 8 weeks
  4 point salivary cortisol is measured over the course of a day
Skin Hydration | 8 weeks
  Delfin MoisturemeterSC 0-150
Facial Redness - Image Based | 8 weeks
  BTBP Clarity Mini 3D camera

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — Integrative Skin Science and Research Institute
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States